CLINICAL TRIAL: NCT07129226
Title: Musculoskeletal Cancers Remote Monitoring and Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CASE1725
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Osteosarcoma; Metastatic Bone Disease
Keywords: prophylactic surgery
MeSH Terms: conditions — Osteosarcoma; Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sarcoma patients (Experimental)
  Interventions: Other: Smart Watch
- Palliative radiation for metastatic bone disease patients (Experimental)
  Interventions: Other: Smart Watch
- prophylactic surgery for metastatic bone disease patients (Experimental)
  Interventions: Other: Smart Watch

INTERVENTIONS:
Other: Smart Watch — Participants will be asked to wear the smartwatch daily, for at least 12 hours per day during the 12-week study period, with breaks to recharge the watch as needed.

SUMMARY:
This study aims to evaluate how walking stability and the ability to perform daily activities change during cancer treatment, and whether a smartwatch can detect these changes. The goal is to develop proactive, personalized tools that automatically monitor treatment response and predict potential complications. To support future implementation, the study will assess the feasibility of wearing a smartwatch for at least 12 hours per day, using a mobile application, and completing weekly questionnaires among patients with primary osteosarcoma or metastatic bone disease.

DETAILED DESCRIPTION:
Wearable sensors, in the form of direct-to-consumer devices, can provide insight to allow timely, proactive, personalized interventions. Nearly 20 percent of US residents own a smart wearable device such as a FitBit or Apple watch. Increasing accessibility and affordability of wearable technology has also allowed for new possibilities to provide personalized and remote care to patients . In part due to the range of sensors in consumer devices that capture multi-modal information. For example, transdermal optical photoplethysmography provides cardiac and respiratory measurements using non-invasive blood flow data. Motion and spatial data are supplied by accelerometers and gyroscopes. These raw data can then be assembled to provide insight into biometric parameters ranging from gait symmetry and step count to higher-level information (e.g. VO2 max and sleep duration).

Our proprietary mobile application (established for Dr. Barker-Clarke's trial NCT06129760 in neurooncology) advances beyond current studies by providing access to raw sensor data and derived mobile health metrics while simultaneously providing a platform for electronic PRO questionnaires. Based on this prior study, investigator anticipate patient eligibility to enroll in this study at around 75% of the patient population, and completed enrollment of around 60% of those eligible. Additionally, having demonstrated the efficacy of our pipeline platform, investigator expects that the collection of ePROMs and actigraphy data will be successful in the patients enrolled. Investigator includes the collection of raw data and derived metrics such as gait asymmetry, breathing rate, and sleep patterns to identify potential digital signatures of recovery, fatigue, or decline that may not be captured by TESS alone. In this new cohort investigator will evaluate compliance in the collection of actigraphy data and reporting of ePROMs. Investigator will estimate effect sizes for actigraphic and gait changes through recovery and anticipate their use in quality of care management or interventional studies in larger patient cohorts. Investigator assume, based on prior studies, that a smartwatch will be able to be worn by at least 80% of the study participants for at least 12 hours per 24-hour period, on average. Investigator outline a study using consumer-grade smartwatches and an application on the patient's phone to collect continuous actigraphy data and ePRO evaluation. In the absence of similar cohort studies for retrospective analysis, investigator aims to generate novel contextualized wearable sensor datasets for musculoskeletal cancer patients and develop digital biomarkers for patient recovery and complications.

ELIGIBILITY:
Inclusion Criteria:

* primary sarcoma or metastatic bone disease of the lower extremities or pelvis.
* undergoing evaluation for radiological or surgical intervention.
* recent Karnofsky Performance Status (KPS) ≥ 70% at baseline.

Exclusion Criteria:

* under 18 years of age at the time of study enrolment
* inability to comprehend consent form and give informed consent
* no access to a smartphone (iOS or Android) to interface with watch application
* tattoos located on the skin of the wrist or forearm where the watch will be placed or other skin conditions preventing adequate sensor function
* amputation or other disease of the arm or skin that prevents wear of a smart-watch device
* inability to tolerate watch for at least 12 hours per day on at least 80% of days in a four-week period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adherence Rate post surgery in patients with sarcoma of the lower extremity or pelvis | 3 months
  Adherence in each case involves averaging ≥ 12h/day wear time and completion in ≥10 out of 12 weeks of the TESS instrument
e-QOL post-surgery in patients with sarcoma of the lower extremity or pelvis | 3 months
Adherence Rate post surgery in patients with metastatic bone disease of the lower extremity or pelvis | 3 months
  Adherence in each case involves averaging ≥ 12h/day wear time and completion in ≥10 out of 12 weeks of the TESS instrument
e-QOL post-surgery in patients with metastatic bone disease of the lower extremity or pelvis | 3 months
Adherence Rate post-radiation in patients with metastatic bone disease of the lower extremity or pelvis | 3 months
  Adherence in each case involves averaging ≥ 12h/day wear time and completion in ≥10 out of 12 weeks of the TESS instrument
e-QOL post-radiation in patients with metastatic bone disease of the lower extremity or pelvis | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No